CLINICAL TRIAL: NCT01779817
Title: Assessment of Intellectual, Psychological and Behavioural Developments Between 6 and 9 Years of the Children Born to Hyperthyroid Mothers During Pregnancy
Brief Title: Assessment of Intellectual, Psychological and Behavioural Developments Between 6 and 9 Years of the Children Born to Hyperthyroid Mothers During Their Pregnancy
Acronym: EDIEMHYPER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PHRC 2011-01
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Hyperthyroid
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- child born to hyperthyroid mother during pregnancy (Other): Assessment of intellectual development, capacities of attention, learning process and degree of hyperactivity of the children between 6 and 9 years.
  Interventions: Behavioral: Assessment of intellectual development, capacities of attention, learning process and degree of hyperactivity of the children between 6 and 9 years.
- child born to euthyroid mother during pregnancy (Other): Assessment of intellectual development, capacities of attention, learning process and degree of hyperactivity of the children between 6 and 9 years.
  Interventions: Behavioral: Assessment of intellectual development, capacities of attention, learning process and degree of hyperactivity of the children between 6 and 9 years.

INTERVENTIONS:
Behavioral: Assessment of intellectual development, capacities of attention, learning process and degree of hyperactivity of the children between 6 and 9 years.

SUMMARY:
1. MAIN OBJECTIVE :

   To assess the consequences of a maternal hyperthyroïd during pregnancy on intellectual development of the child from 6 to 9 years
2. SECONDARY OBJECTIVES :

   1. To assess the consequences of a maternal hyperthyroïd during pregnancy on the capacities of attention, learning process and the degree of hyperactivity of the child from 6 to 9 years.
   2. To study if it exist differences of intellectual development, capacities of attention, learning process, and degree of hyperactivity in the child from 6 to 9 years, born to hyperthyroid mother during pregnancy, according to:

      * the etiology of the maternal hyperthyroïd (transitory gestation hyperthyroid versus disease of Basedow),
      * the use or not of a anti-thyroid treatment,
      * the rate of TSH néonatal (measured with the blotter by tracking with J3 at all the new born ones).

DETAILED DESCRIPTION:
1. INCLUSION CRITERIA :

   * Old from 6 to 9 years included
   * Age of gestation between ≥37 and <41 weeks of amenorrhoea
   * Born from a mono-foetale pregnancy
   * Euthyroïd at the time of the entry in the study
   * Provided education for at the elementary school on a level adapted to its age
2. NON INCLUSION CRITERIA :

   * Presenting a congenital hypothyroïd or a known thyroid dysfonction at the time of the entry in the study
   * Carrier of a chronic pathology (organic or psychological) or malformative severe
   * Presenting an antecedent of Deficit of the Attention-Hyperactivity to the 1st degree
3. EXCLUSION CRITERIA :

   o Discovered of a thyroid dysfonction at the time of the entry in the study
4. STRATEGIES / PROCEDURES :

Multicentric, comparative study of a troop of child born to hyperthyroïd mothers during pregnancy (children exposed to the maternal hyperthyroïd) and children born to euthyroïd mothers during pregnancy (nonexposed children with the maternal hyperthyroïd).

* 1st part of the study: Retrospective analyze of the files of symptomatic hyperthyroid mothers during pregnancy.
* 2nd part of the study: Assessment of intellectual development, capacities of attention, learning process and degree of hyperactivity of the children between 6 and 9 years. The exposed children (born to hyperthyroïd mothers during pregnancy) will be compared with nonexposed children (born to euthyroïd mothers during pregnancy).

ELIGIBILITY:
1. Inclusion Criteria:

   A-For the child born to hyperthyroid mother during pregnancy :

   oOld from 6 to 9 years included oAge of gestation between ≥37 and <41 weeks of amenorrhoea oBorn from a mono-foetale pregnancy oEuthyroïd at the time of the entry in the study oProvided education for at the elementary school on a level adapted to its age

   B-For hyperthyroid mother during pregnancy :

   oHyperthyroïd during pregnancy (transitory gestation hyperthyroid or disease of Basedow) oEuthyroïd at the time of the entry in the study

   C-For the child born to euthyroid mother during pregnancy :

   oOld from 6 to 9 years included oAge of gestation between ≥37 and <41 weeks of amenorrhoea oBorn from a mono-foetale pregnancy oEuthyroïd at the time of the entry in the study oProvided education for at the elementary school on a level adapted to its age

   D-For euthyroid mother during pregnancy :

   Euthyroïd at the time of the entry in the study
2. Exclusion Criteria:

A-For the child born to hyperthyroid mother during pregnancy :

Discovered of a thyroid dysfonction at the time of the entry in the study

B-For hyperthyroid mother during pregnancy:

Discovered of a thyroid dysfonction at the time of the entry in the study

C-For the child born to euthyroid mother during pregnancy:

Discovered of a thyroid dysfonction at the time of the entry in the study

D-For euthyroid mother during pregnancy:

oDiscovered of a thyroid dysfonction at the time of the entry in the study oCarrying anti-TPO antibody at the time of the entry in the study

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 252 (Estimated)
Dates: Start 2013-02; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Scores of global development Quotient (WISC-R) | within the first 30 days after inclusion of the patient

SECONDARY OUTCOMES:
Score of the Achenbach Child Behavior Checklist | within the first 30 days after inclusion of the patient
Score of the conners scale | within the first 30 days after inclusion of the patient
Score of the Wechsler Intelligence Scale for Children (WISC-IV) | within the first 30 days after inclusion of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Natacha BOUHOURS-NOUET, Principal Investigator — UNIVERSITY HOSPITAL OF ANGERS
Locations (13):
- France (13):
  - University Hospital of Amiens, Amiens
  - University Hospital of Angers, Angers
  - Civil Hospices of Lyon, Bron
  - University Hospital of Kremlin Bicetre, Le Kremlin-Bicêtre
  - University Hospital of Lille, Lille
  - University Hospital of Marseille, Marseille
  - University Hospital of Nantes, Nantes
  - Hospital of Saint Antoine, Paris
  - University Hospital of Cochin, Paris
  - University Hospital of Poitiers, Poitiers
  - University Hospital of Reims, Reims
  - University Hospital of Strasbourg, Strasbourg
  - University Hospital of Toulouse, Toulouse